CLINICAL TRIAL: NCT00016458
Title: Phase II Pilot Study of Cyclophosphamide and Rabbit Anti-Thymocyte Globulin as Salvage Therapy in Patients With Diffuse Systemic Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/15818; FHCRC-1473.00
Record Dates: First submitted 2001-05-06; First posted 2001-05-07 (Estimated); Last update posted 2008-09-03 (Estimated); Status verified 2008-09

CONDITIONS: Systemic Sclerosis
Keywords: arthritis & connective tissue diseases; rare disease; systemic sclerosis
MeSH Terms: conditions — Scleroderma, Systemic; Arthritis; Connective Tissue Diseases; Rare Diseases | interventions — Antilymphocyte Serum; Cyclophosphamide

INTERVENTIONS:
Drug: anti-thymocyte globulin
Drug: cyclophosphamide

SUMMARY:
OBJECTIVES: I. Determine the toxicity of cyclophosphamide and rabbit anti-thymocyte globulin in patients with diffuse systemic sclerosis.

II. Determine the efficacy of this regimen in terms of controlling disease in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients receive cyclophosphamide IV over 1-2 hours on day 1 and rabbit anti-thymocyte globulin IV over 6-8 hours on days 2-5.

Patients are followed on days 60-85 and then every 3 months for 1 year.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Diagnosis of diffuse systemic sclerosis

Progressive disease Skin score at least 16 Interstitial or pulmonary vasculitis (FVC or DLCO no greater than 70% predicted) with evidence of alveolitis by bronchoalveolar lavage (BAL) Proteinuria (more than 500 mg/24 hours) Rapid deterioration in pulmonary function (at least 15% decrease in FVC or DLCO within the past 6 months) or new evidence of alveolitis by CT scan changes or BAL

No acute renal failure secondary to systemic sclerosis crisis

DLCO greater than 20% predicted

Ineligible for or refused autologous or allogeneic peripheral blood stem cell or bone marrow transplantation

--Prior/Concurrent Therapy--

Endocrine therapy: Concurrent prednisone allowed if prior chronic use

Other: At least 4 days since prior immunosuppressive therapy

--Patient Characteristics--

Performance status: Karnofsky 50-100%

Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3

Hepatic: Bilirubin less than 2.5 times upper limit of normal (ULN) SGOT less than 2.5 times ULN

Renal: See Disease Characteristics Creatinine clearance at least 35 mL/min No requirement for renal dialysis

Cardiovascular: Ejection fraction greater than 45% No myocardial infarction within the past 12 months No unstable angina No uncontrolled cardiac arrhythmias No evidence of congestive heart failure

Pulmonary: See Disease Characteristics

Other:

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No active uncontrolled infection
* No hypersensitivity to rabbit proteins
* No prior hemorrhagic cystitis requiring transfusion
* No concurrent active hemorrhagic cystitis by cystoscopy (if prior history)
* No concurrent malignancy

Max Age: 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20
Dates: Start 2000-06

CONTACTS AND LOCATIONS:
Overall Officials: Leona Holmberg, Study Chair — Fred Hutchinson Cancer Center
Locations (3):
- United States (3):
  - University of Colorado Cancer Center, Denver, Colorado
  - Duke University Medical Center, Durham, North Carolina
  - Fred Hutchinson Cancer Research Center, Seattle, Washington